CLINICAL TRIAL: NCT06528470
Title: A Randomized Controlled Trial of Posterior Tibial Nerve Stimulation for Children With Constipation Due to Pelvic Floor Dyssynergia
Brief Title: Posterior Tibial Nerve Stimulation for Children With Pelvic Floor Dyssynergia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Peter Lu, Pediatric Gastroenterologist, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000403
Record Dates: First submitted 2020-09-11; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Constipation; Fecal Incontinence in Children; Pelvic Floor Dyssynergia
Keywords: Posterior Tibial Nerve Stimulation; Neuromodulation; Constipation; Fecal Incontinence; Pelvic Floor Dyssynergia; Children
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Posterior Tibial Nerve Stimulation (PTNS) (Experimental): Patients in the PTNS arm will undergo 30-minute sessions of PTNS after their first four pelvic floor biofeedback therapy sessions.
  Interventions: Device: Posterior Tibial Nerve Stimulation (PTNS)
- Sham Stimulation (Sham Comparator): Patients in the PTNS arm will undergo 30-minute sessions of sham stimulation after their first four pelvic floor biofeedback therapy sessions.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Posterior Tibial Nerve Stimulation (PTNS) — The intervention will begin with application of a needle and a self-adhesive electrode. The electrodes will be connected to the electrical stimulator device. The stimulator will then be turned on and amplitude will be gradually increased until motor or sensory response is observed. The amplitude will then be decreased to the point when direct motor stimulation ceases and sensory stimulation is comfortable. Continuous stimulation will then be delivered for a 30-minute session. After 30 minutes, the device will be turned off and the adhesive electrodes removed. Pelvic floor biofeedback therapy is typically performed for a total of four or more weekly sessions. Participants in our study will undergo 30-minute sessions of PTNS or sham stimulation after their first four biofeedback therapy sessions.
  Other Names: Urgent PC (Cogentix Medical, Minnetonka, MN)
  Arms: Posterior Tibial Nerve Stimulation (PTNS)
Device: Sham Stimulation — The intervention will begin with application of a needle and a self-adhesive electrode. The electrodes will be connected to the electrical stimulator device. The stimulator will then be turned on and amplitude will be gradually increased until motor or sensory response is observed. The amplitude will then be decreased to the point when no stimulation is delivered. No stimulation will then be delivered for a 30-minute session. After 30 minutes, the device will be turned off and the adhesive electrodes removed. Pelvic floor biofeedback therapy is typically performed for a total of four or more weekly sessions. Participants in our study will undergo 30-minute sessions of PTNS or sham stimulation after their first four biofeedback therapy sessions.
  Other Names: Urgent PC (Cogentix Medical, Minnetonka, MN)
  Arms: Sham Stimulation

SUMMARY:
The overall objective of this study is to determine the effect of posterior tibial nerve stimulation (PTNS) on children with constipation due to pelvic floor dyssynergia. Our main hypothesis is that PTNS effectively treats children with constipation secondary to pelvic floor dyssynergia through modulation of anorectal function. We will perform a single-center, randomized controlled pilot study comparing PTNS to sham stimulation in children with constipation secondary to pelvic floor dyssynergia.

DETAILED DESCRIPTION:
Constipation affects up to 30% of children in population-based studies and 15% of children with constipation will continue to have symptoms despite years of aggressive medical treatment. Pelvic floor dyssynergia, which involves abnormal coordination of pelvic floor muscles during defecation, is a common finding during anorectal manometry testing for children with refractory constipation. Treatment options for children with constipation refractory to medical treatment are limited and generally invasive. Thus, there is an urgent need for the identification and evaluation of non-invasive treatments for constipation refractory to medical treatment. We have established, through research at our institution, that electrical stimulation delivered via gastric electrical stimulator and sacral nerve stimulator is feasible and effective in the treatment of gastrointestinal disease. There is new evidence that posterior tibial nerve stimulation (PTNS), a non-invasive method of delivering electrical stimulation, can be effective in the treatment of adults with constipation and fecal incontinence. Our long-term goal is to identify and evaluate novel non-invasive treatment options for children with constipation refractory to medical treatment.

The overall objective of this study is to determine the effect of PTNS on children with constipation due to pelvic floor dyssynergia. Our main hypothesis is that PTNS effectively treats children with constipation secondary to pelvic floor dyssynergia through modulation of anorectal function. We plan to objectively test our main hypothesis and attain the objective of this application by pursuing the following specific aims:

AIM 1: Determine the efficacy of PTNS in the treatment of children with constipation due to pelvic floor dyssynergia. The working hypothesis is that PTNS will lead to improvement in validated measures of constipation severity.

AIM 2: Determine the effects of PTNS on anorectal function. The working hypothesis is that PTNS will lead to improvement in pelvic floor dyssynergia.

The expected outcome of Aim 1 is demonstration that PTNS is effective in decreasing the symptom severity of children with constipation due to pelvic floor dyssynergia. Aim 2 will show that PTNS improves symptoms by modulating anorectal function. Establishing that PTNS is an effective treatment option for children with constipation due to pelvic floor dyssynergia will have a significant positive impact on a population of children for which management is challenging and current therapeutic options are limited. Determining the mechanism by which PTNS acts will further our understanding of the effect of electrical stimulation on the human body and could lead to identification of other applications of therapeutic electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 8-18 years of age
* Diagnosis of constipation due to pelvic floor dyssynergia
* Scheduled to start pelvic floor biofeedback therapy.

Exclusion Criteria:

- Prior surgery for constipation (colonic resection, cecostomy, Malone appendicostomy, sacral nerve stimulator implantation, etc.)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Cleveland Clinic Constipation Score (CCCS) | 4 weeks after starting treatment
  We will use the Cleveland Clinic Constipation Score (CCCS) to measure constipation severity.
Fecal Incontinence Severity Index (FISI) | 4 weeks after starting treatment
  We will use the Fecal Incontinence Severity Index (FISI) to measure fecal incontinence severity.

SECONDARY OUTCOMES:
Cleveland Clinic Constipation Score (CCCS) | 5 weeks after starting treatment
  We will use the Cleveland Clinic Constipation Score (CCCS) to measure constipation severity.
Cleveland Clinic Constipation Score (CCCS) | 8 weeks after starting treatment
  We will use the Cleveland Clinic Constipation Score (CCCS) to measure constipation severity.
Fecal Incontinence Severity Index (FISI) | 5 weeks after starting treatment
  We will use the Fecal Incontinence Severity Index (FISI) to measure fecal incontinence severity.
Fecal Incontinence Severity Index (FISI) | 8 weeks after starting treatment
  We will use the Fecal Incontinence Severity Index (FISI) to measure fecal incontinence severity.

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Lu, MD, MS, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No